CLINICAL TRIAL: NCT06643286
Title: Personalised Survivorship Care for Patients With Melanoma: A Multicenter Randomised Controlled Trial of the Survivorship Care Plan App
Brief Title: Evaluation of a Personalised Survivorship Care Plan App for Patients With Melanoma
Acronym: Melanoma SCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: BeterKeten (Unknown); Albert Schweitzer Hospital (Other); Maasstad Hospital (Other); Franciscus Gasthuis (Other)
Responsible Party: Principal Investigator, Marjolein Lugtenberg, Doctor, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 10147
Record Dates: First submitted 2024-10-08; First posted 2024-10-16 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-04

CONDITIONS: Melanoma (Skin); Melanoma, Stage II, Stage I; Melanoma Stage; Survivorship
Keywords: Survivorship care; Application; RCT
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: Multicentre randomized controlled trial, in which participants are randomised to either the intervention group (use of the intervention in addtion to care usual) or the control group (solely care as usual).
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care as usual is not altered in both study groups, as to where the care providers continue to deliver the same care. As they are unaware of availability of the intervention, the degree of information provision is not compromised.
  During quantitative analyses we pursue masking the outcomes assessor(s).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants receive access to the Digizorg Melanoma app, on top of care as usual.
  Interventions: Device: Digizorg Melanoma app
- Control group (No Intervention): Participants have access to care as usual, but have no access to the Digizorg Melanoma app and its functionalities.

INTERVENTIONS:
Device: Digizorg Melanoma app — The Digizorg Melanoma app is a digital survivorship care plan, in which ellaborated information regarding diagnosis, treatment and follow-up and supportive care, adjusted to one's personal preferences and disease characteristics, is offered in the form of a mobile application.
  Arms: Intervention group

SUMMARY:
A multicentre randomised controlled trial (RCT) will be conducted to evaluate the effectiveness of the digital personalised Melanoma Survivorship Care Plan (SCP) app. A total of hundred-eighty melanoma patients (stage I and II) will be randomised to receive either the SCP Melanoma app or usual care. The app provides survivors with personalized healthcare information on diagnosis, treatment and follow-up and supportive care, tailored to their melanoma stage and phase and information needs.Through questionnaires, medical file records, patient-reported outcomes and use of medical care will be evaluated. In addition, log-data, questionnaires and interviews will be used to evaluate the process of the uptake and implementation of the digital SCP.

DETAILED DESCRIPTION:
The growing and diverse group of survivors of stage I and II melanoma leads to an increasing need for patient-tailored survivorship care. To meet these needs, the Survivorship Care Plan (SCP) app ('Digizorg Melanoma app') was developed together with patients and healthcare providers, providing patients with melanoma with personalised information on diagnosis, treatment and follow-up and supportive care. The aim of this study is to evaluate the effectiveness of the Digizorg Melanoma SCP app in terms of patient and provider-reported outcomes and clinical practice.

A multicenter randomized controlled trial (RCT) will be performed in four Dutch hospitals, namely Erasmus MC, Albert Schweitzer hospital, Maasstad hospital and Franciscus Gasthuis & Vlietland. A total of 180 patients (stage I and II) will be randomized to receive either the 'SCP-app' or 'usual care'. Patients are included within 0-4 months of primary diagnosis. If patients are diagnosed with stage III or IV, they are excluded. The app consists of information tailored to survivors' melanoma stage and phase as well as their information needs. Participants receive questionnaires at baseline, and at 6 and 12 months. Additionally, medical records are examined for healthcare use. The primary outcome is patient empowerment. Secondary outcomes are satisfaction with information and care, fear of (return of) cancer, needs for supportive care, coping style and healthcare use. Additionally, a process evaluation will be conducted to gain insight into the uptake and evaluation of (the implementation of) the intervention by users.

To evaluate the effectiveness of the Digizorg Melanoma app (effect evaluation), scores on outcome measures will be compared between the two study groups through questionnaires and medical file records analysis, correcting for baseline scores. The primary outcome measure is patient empowerment. Secondary outcome measures are medical care consumption, costs, fear of (return of) cancer, need for supportive care, coping style and satisfaction with information and care. All outcome measures are measured in both groups in the form of questionnaires at the start of the trial (T0) and 6 (T1) and 12 months (T2) after inclusion. Medical file records (number of healthare appointment records in the file) will only be assessed at the start of the trial (T0) and after 12 months (T2).

To gain insight into the uptake and evaluation of (the implementation of) the intervention (process evaluation), (log) data on the use of the app will be analysed, short satisfaction questionnaires will be administered twice to patients and up to 30 short-term interviews with patients and other stakeholders (including healthcare providers, IT specialists and developers) will be conducted to explore satisfaction with app, impact on coordination and suggestions for improvement.

There are no specific risks associated with participating in this study. Participants will have the opportunity to use the app with personalised information on diagnosis, treatment and follow-up and supportive care. However, no specific actions are imposed and the care participants receive remains the same. Participation in the study does require a time investment from patients in the form of completing questionnaires three times over a year. However, the time investment will be limited to 30-45 minutes each time. In addition, the number of questions that can be perceived as burdensome by patients is limited. A small proportion of patients will additionally be approached for a short-term interview (of max 30 min) as part of the process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients who have received a primary diagnosis of cutaneous melanoma stage I to II in the past 0-4 months

Exclusion Criteria:

* Patients with irresectable stage III melanoma, patients receiving neo-adjuvant treatment and patients with stage IV melanoma.
* Patients who do not have (sufficient) command of the Dutch language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient empowerment | 1 year after inclusion
  The extent to which patients are able to cope with their own condition. This is a result of understanding by the patient of his/her role, acquisition by patients of sufficient knowledge to be able to engage with their healthcare provider, the skills of the patient skills and the presence of a facilitating environment. This outcome is measured through a scaled questionnaire (Health Education Impact Questionnaire), on which higher scores indicate a more health-conscious, self-monitored and empowered self.

SECONDARY OUTCOMES:
Medical care consumption | 1 year after inclusion
  The amount of (additional) contact moments (including telephone consultations) with medical specialists, nursing specialists and assistant physicians in the hospital, on top of care as usual.This outcome is measured in volumina through a questionnaire (iMTA Medical Consumption Questionnaire) and medical file research.
Costs | 1 year after inclusion
  All medical costs, related to healthcare utilization, and non-medical costs, related to productivity loss and implementation of the application. This outcome is calculated through the volumes of medical care consumption and productivity loss.
Satisfaction with care | 1 year after inclusion
  Overall subjective assessment of the received care around melanoma. This outcome is measured through one scaled question of a questionnaire (EORTC Outpatient satisfaction 7-items), of which lower scores indicate less satisfaction with care.
Fear of recurrence | 1 year after inclusion
  The extent of worries and fears surrounding cancer in oncology patients. This outcome is measured through a questionnaire (Cancer Worry Scale). Higher scores indicate more distress around cancer recurrences.
Coping style | At baseline
  The thoughts and behaviors mobilized to manage internal and external stressful situations. This outcome is measured through a questionnaire (shortened Threatening Medical Situations Inventory), in which two hypothetical situations and resulting actions are assessed and scored.
Productivity loss | 1 year after inclusion
  The extent to which the person's ability to perform his/her work is affected as a result of the disease. This outcome is measured in volumina through a questionnaire (iMTA productivity cost questionnaire).
Satisfaction with information | 1 year after inclusion
  The extent and quality to which patients feel informed, specifically during treatment for melanoma. This outcome is measured through a questionnaire (EORT Core Quality of Life Questionnaire Information module 25-items), by which self-report can express high satisfaction with information (high scores) to low satisfaction (low scores).
Need for supportive care | 1 year after inclusion
  The individual needs of the patient for care, upon which targeted supportive care can then be provided. This outcome is measured through a questionnaire (Supportive Care Needs Survey - Short form 34-items), exposing different areas for needs through distinguishment of the level of satisfaction and need for care.

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Albert Schweitzer hospital, Dordrecht, South Holland
  - Erasmus MC, Rotterdam, South Holland
  - Franciscus Gasthuis & Vlietland hospital, Rotterdam, South Holland
  - Maasstad hospital, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Undecided